CLINICAL TRIAL: NCT06170983
Title: Validation of Imiquimod- and LPS-induced Skin Inflammation Models and Their Application in the Investigation of Azithromycin Concentration in Inflamed, Infected, and Healthy Subcutaneous Tissue
Brief Title: Skin Inflammation and PK of Azithromycin
Acronym: AZI_IMQ_LPS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Markus Zeitlinger, MD, Medical University of Vienna
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: Pro_AZI_IMQ_LPS
Record Dates: First submitted 2023-11-27; First posted 2023-12-14 (Actual); Last update posted 2023-12-14 (Actual); Status verified 2023-12

CONDITIONS: Skin Infection
MeSH Terms: conditions — Cellulitis | interventions — Azithromycin; Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Pilot Cohort for Skin Inflammation (Experimental): Testing skin inflammation
  Interventions: Diagnostic Test: Biopsy; Other: Skin inflammation model
- Azithromycin and Artificial Skin Inflammation (Experimental): Investigating tissue PK of Azithromycin in artificially inflamed tissue
  Interventions: Drug: Azithromycin; Other: Skin inflammation model
- Azithromycin and Skin Infection (Experimental): Investigating tissue PK of Azithromycin in actually infected tissue
  Interventions: Drug: Azithromycin

INTERVENTIONS:
Drug: Azithromycin — 500 mg once daily for 3 days
  Arms: Azithromycin and Artificial Skin Inflammation; Azithromycin and Skin Infection
Diagnostic Test: Biopsy — Skin punch biopsy
  Arms: Pilot Cohort for Skin Inflammation
Other: Skin inflammation model — LPS- or imiquimod induced skin inflammation
  Arms: Azithromycin and Artificial Skin Inflammation; Pilot Cohort for Skin Inflammation

SUMMARY:
This study will investigate the tissue distribution of azithromycin in healthy, artificially inflamed and actually infected tissue of humans.

DETAILED DESCRIPTION:
This single-center, prospective, open-label, adaptive, pharmacokinetic study will comprise three parts: Part 0a-c, Part A, and Part B.

Objectives: This study primarily aims to characterize and establish a new skin inflammation model using topically applied LPS. The secondary aim of this research is to deepen our understanding of the role of leukocytes as potential transport vehicles for macrolides and other antibiotics in humans.

Intervention: Part 0 will serve as a pilot experiment in healthy volunteers to validate the imiquimod and LPS challenge in a controlled design. The investigators will clinically assess the tolerability of increasing LPS doses and the already published design of the imiquimod challenge. In general, the investigators will perform the different designs of skin inflammation models using tape stripping and an occlusive 18-mm Finn chamber.

The inflammation will not only be clinically assessed but also objectively quantified using the imaging-based mobile phone application Scarletred®Vision. Considering these results, the investigators will again carry out the LPS and imiquimod challenge in healthy volunteers and additionally perform biopsies in Part 0c to collect specimens for flow cytometry. Thus, the investigators will be able to characterize the skin inflammation models at a cellular level. Using NGS, the investigators will also explore transcriptional changes within cell subset that are affected by the inflammation.

In Part 0c, the investigators will include 12 healthy volunteers and will perform in each subject three skin punch biopsies, including a negative control, IMQ-challenged skin and LPS-challenged skin. Using flow cytometry, the investigators will measure the infiltration of leukocytes subsets.

Part A will employ a skin inflammation challenge based on either LPS or the imiquimod according to the results of Part 0 (i.e., the one showing the greater leucocyte infiltration). Azithromycin will be given in parallel once daily for 3 consecutive days. After the last application (i.e. day 3), two microdialysis probes will be placed in the inflamed subcutaneous tissue and one will be placed in the unmanipulated healthy subcutaneous fat. Hereafter, PK sampling and microdialysis of two thighs will be performed for two consecutive days. The investigators will isolate leukocytes from blood samples on day 3 to determine the average concentration of azithromycin in them. Biopsies from the unmanipulated and the challenged skin will be obtained on day 4.

Part B will involve patients with skin infections including erysipelas and cellulitis at their lower extremities. In contrast to Part A, only one microdialysis probe will be placed into the infected subcutaneous tissue and one into healthy, unaffected tissue. After three doses of azithromycin, pharmacokinetic sampling, leukocyte isolation, and microdialysis of the healthy thigh and the respective area of infection will be performed.

ELIGIBILITY:
Inclusion Criteria:

* • Men and women aged ≥18 and <55 years

  * BMI ≥18 and ≤30 kg/m2
  * Normal (or clinically irrelevant abnormal) findings in medical history and physical examination
  * Women with child-bearing potential: use of effective contraception
  * Laboratory parameters within the given reference range (or abnormal findings which are irrelevant for study purposes in the Investigator's opinion)

Exclusion Criteria:

* Known or suspected allergy to lipopolysaccharide, imiquimod, or sticking plasters
* Only Part 0c: Known or suspected allergy to local anesthetics
* History of severe allergic or anaphylactic reactions to any medication • Blood donation within the last 4 weeks before the study
* Treatment with an investigational drug within three weeks before the study
* Smoking of more than 5 cigarettes per day
* Regular use of medication or abuse of alcohol
* Use of any medication within one week before the study
* Symptoms of a clinically relevant illness in the 3 months before the study
* Liver or kidney dysfunction
* Pregnancy
* History of autoimmune diseases (especially psoriasis)
* Other objections to participating in the study in the opinion of the Investigator

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Part 0: Area under the curve (AUC) of azithromycin in artificially inflamed tissue | Day 3
  The pharmacokinetic concentration-time profile in tissue will be assessed by microdialysis. Concentration-time profiles will be plotted. AUC and Cmax will be used as PK parameters.
Part 0: Maximum concentration (Cmax) of azithromycin in artificially inflamed tissue | Day 3
  The pharmacokinetic concentration-time profile in tissue will be assessed by microdialysis. Concentration-time profiles will be plotted. AUC and Cmax will be used as PK parameters.
Part A: Area under the curve (AUC) Azithromycin in healthy and inflamed tissue | Day 3
  The pharmacokinetic concentration-time profile in tissue will be assessed by microdialysis. Concentration-time profiles will be plotted. AUC and Cmax will be used as PK parameters.
Part A: Maximum concentration (Cmax) Azithromycin in healthy and inflamed tissue | Day 3
  The pharmacokinetic concentration-time profile in tissue will be assessed by microdialysis. Concentration-time profiles will be plotted. AUC and Cmax will be used as PK parameters.
Part B: Area under the curve (AUC) of Azithromycin in healthy and infected tissue | Day 3
  The pharmacokinetic concentration-time profile in tissue will be assessed by microdialysis. Concentration-time profiles will be plotted. AUC and Cmax will be used as PK parameters.
Part B: Maximum concentration (Cmax) of Azithromycin in healthy and infected tissue | Day 3
  The pharmacokinetic concentration-time profile in tissue will be assessed by microdialysis. Concentration-time profiles will be plotted. AUC and Cmax will be used as PK parameters.

SECONDARY OUTCOMES:
Part 0-A: Safety and tolerability of inflammation models | Day 0-3
  Data will be aggregated as:
  * number of participants with treatment-related local adverse events due to the inflammation models
  * number of participants with treatment-related systemic adverse events due to the inflammation models
Part A-B: Safety and tolerability of azithromycin | Day 0-3
  Data will be presented as:
  * number of participants with treatment-related systemic adverse events due to azithromycin
  * mean number of treatment-related systemic adverse events due to azithromycin per subject

IPD SHARING:
Plan to Share IPD: Undecided